CLINICAL TRIAL: NCT01990859
Title: Phase 2 Study of Ipilimumab in Japanese Subjects With Unresectable or Metastatic Melanoma
Brief Title: Phase 2 Study of Ipilimumab in Japanese Advanced Melanoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-396
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A: Ipilimumab (Experimental): Ipilimumab Intravenous Injection 3 mg/kg for every 3 weeks upto 4 doses
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab
  Other Names: BMS-734016

SUMMARY:
The purpose of this study is to assess the safety of Ipilimumab monotherapy in Japanese subjects with advanced melanoma

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of malignant melanoma
* Previously-treated or untreated unresectable Stage III or Stage IV melanoma
* Measurable/evaluable disease per modified World Health Organization (mWHO) criteria, within 28 days of first dose of study drug
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Active brain metastases
* Primary ocular or mucosal melanoma
* History of or current active autoimmune disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- Japan (6):
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Matsumoto-shi, Nagano
  - Local Institution, Sunto-gun, Shizuoka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Chuo-shi, Yamanashi

REFERENCES:
- [Derived] Yamazaki N, Kiyohara Y, Uhara H, Fukushima S, Uchi H, Shibagaki N, Tsutsumida A, Yoshikawa S, Okuyama R, Ito Y, Tokudome T. Phase II study of ipilimumab monotherapy in Japanese patients with advanced melanoma. Cancer Chemother Pharmacol. 2015 Nov;76(5):997-1004. doi: 10.1007/s00280-015-2873-x. Epub 2015 Sep 26. PMID 26410424
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated 12 December 2013 and completed February 2015. Previously treated or untreated patients with Stage III (unresectable) or Stage IV melanoma were recruited. Previously untreated defined as: patients without treatment for metastatic disease but who may have received treatment in the adjuvant setting.
Pre-assignment Details: 26 participants were enrolled and 20 were treated with study drug. Of the 6 participants not treated: 5 no longer met study criteria, 1 withdrew consent.
Groups:
- Ipilimumab: During treatment, participants received Ipilimumab intravenous (IV) injection 3 mg/kg every 3 weeks, up to 4 doses (12 weeks). Study was divided into 4 Phases: Screening Phase, Induction Phase, Toxicity/Progressive Disease(PD) Follow Up Phase, and Overall Survival Phase. The Induction Phase consisted of treatment and a 12 week post dosing follow up. It started at first dose and ended at Week 24, or earlier if participant discontinued treatment and moved to Follow-Up Phase.
Period: Treatment (4 Doses Over 12 Weeks)
Arm/Group | Ipilimumab
Started | 20
Completed | 15
Not Completed | 5
Not completed — Progressive Disease | 5
Period: Week 12 to Week 24 Post Dosing Follow Up
Arm/Group | Ipilimumab
Started | 20 (All were entered into follow-up whether dosing was completed or not.)
Completed | 3
Not Completed | 17
Not completed — Disease Progression | 17
Period: 90 Day Follow Up for All Participants
Arm/Group | Ipilimumab
Started | 20 (All entered into 90 day follow-up whether treatment and/or post dose follow up was completed or not.)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants in the study who received at least one dose of treatment with ipilimumab were summarized.
Groups:
- Ipilimumab: Participants received Ipilimumab intravenous (IV) injection 3 mg/kg every 3 weeks, up to 4 doses.
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 62.5 [29.0 to 76.0]
Age, Customized [Number; unit: participants]
  Less than 65 years | 13
  Greater than, equal to 65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 20
Region of Enrollment [Number; unit: participants]
  Japan | 20
M-Stage at Study Entry [Number; unit: participants] — Melanoma Tumor Staging: Metastasis (M) classification (M1a versus M1b versus M1c). M1a: Distant skin, subcutaneous tissue, or nodal metastases with normal lactic dehydrogenase (LDH); M1b: Lung metastases with normal LDH; M1c: All other visceral metastases with normal LDH; Any distant metastasis with elevated LDH. Final Version of the American Joint Committee on Cancer Staging System for Cutaneous melanoma. Journal of Clinical Oncology, 2001. (Vol. 19 No.16): p. 3635-3648.
  participants
    M0 | 1
    M1A | 1
    M1B | 4
    M1C | 14
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants] — ECOG PS, is a 6-item scale to assess disease progression, daily functioning, and appropriate treatment and prognosis. Scale: 0-5 with 0=Fully active; 1= restricted in physically strenuous activity; 2= ambulatory; 3=limited self care; 4= completely disabled; 5=dead.
  participants
    ECOG PS 0 | 14
    ECOG PS 1 | 6
Height in centimeters (cm) [Median (Full Range); unit: cm] | 161.7 [144.0 to 184.6]
Weight in kilograms (kg) [Median (Full Range); unit: kg] | 64.0 [40.8 to 109.0]
Baseline Lactate Dehydrogenase (LDH) [Number; unit: participants] — Elevation defined as greater than (>) Upper Limit of Normal (ULN) limit.
  participants
    Normal | 8
    Elevated | 12
Baseline LDH Greater than 2 Times Upper Limit of Normal [Number; unit: participants] — Elevation in this baseline characteristic was defined as greater than (>) 2 Times the Upper Limit of Normal
  participants
    Normal | 13
    Elevated | 7
Prior Systemic Anti-Cancer Therapy [Number; unit: participants]
  Yes | 16
  No | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation of Study Drug, Related AEs, Immune-related AEs (IrAEs) at Primary Endpoint - All Treated Participants
Description: AEs graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death. Related=relationship to study drug reported as certain, probable, possible, or missing. Immune-related AEs (irAEs) characterized by potential association with inflammation and considered by investigator as drug related. Primary endpoint (PE) includes results from Day 1 to 12 weeks after initial dose of last participant. Data evaluated at PE last patient, last visit (LPLV).
Time Frame: Day 1 to 90 Days after the last dose, up to May 2014
Population: All participants in the study who received at least one dose of treatment with ipilimumab were summarized. Data up to May 2014 included.
Measure: Number; unit: participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
participants
  Deaths | 6
  Deaths Due to Disease Progression | 6
  SAEs | 10
  Treatment-Related SAEs | 3
  AEs Leading to Discontinuation of Study Drug | 1
  Grade 3/4 AEs | 7
  Treatment-Related AEs | 12
  Grade 3/4 Related AEs | 3
  irAEs | 12
  Grade 3/4 irAEs | 2

2. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation of Study Drug, Related AEs, Immune-related AEs (IrAEs) - All Treated Participants
Description: AEs graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death. Related=relationship to study drug reported as certain, probable, possible, or missing. Immune-related AEs (irAEs) characterized by potential association with inflammation and considered by investigator as drug related.
Time Frame: Day 1 to 90 Days after the last dose, up to July 2014
Population: All participants in the study who received at least one dose of treatment with ipilimumab were summarized.
Measure: Number; unit: participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
participants
  Deaths | 8
  Deaths Due to Disease Progression | 8
  SAEs | 11
  Treatment-Related SAEs | 3
  AEs Leading to Discontinuation of Study Drug | 1
  Grade 3/4 AEs | 9
  Treatment-Related AEs | 12
  Grade 3/4 Related AEs | 3
  irAEs | 12
  Grade 3/4 irAEs | 3

3. Secondary Outcome: Number of Participants Who Died - All Treated Participants
Description: Total number of deaths that occurred in all treated participants by study completion are reported.
Time Frame: Day 1 to 90 days post last dose, up to February 2015 (approximately 2 years)
Population: All participants in the study who received at least one dose of treatment with ipilimumab were summarized.
Measure: Number; unit: participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
participants
  Deaths within 90 days of last dose | 5
  Deaths at greater than 90 days post last dose | 8

4. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities
Description: Abnormal laboratory results were reported after the induction period start and within 90 days after induction period end date. Induction Period was 1 dose every 3 weeks for 4 doses (12 weeks). Common Terminology Criteria (CTC) version 3.0 was used in this study; Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death. Hematology parameters included: White Blood Cell Count (WBC), Absolute Neutrophil Count, Platelet Count, Hemoglobin, and Lymphocyte Count (absolute). The most recent assessment on or before Day 1 of study medication was taken as baseline (in addition, baseline laboratory must have been collected no earlier than Day -28).
Time Frame: Baseline to 90 days post last dose, up to July 2014
Population: All participants in the study who received at least one dose of treatment with ipilimumab and had laboratory data were summarized. Data included up to July 2014.
Measure: Number; unit: participants
Groups:
- Ipilimumab: During treatment, participants received Ipilimumab IV injection 3 mg/kg every 3 weeks, up to 4 doses (12 weeks). Study was divided into 4 Phases: Screening Phase, Induction Phase, Toxicity/Progressive Disease (PD) Follow Up Phase, and Overall Survival Phase. The Induction Phase consisted of treatment and a 12 week post dosing follow up. It started at first dose and ended at Week 24, or earlier if participant discontinued treatment and moved to Follow-Up Phase.
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
participants
  WBC Grade 1-4 | 1
  WBC Grade 3-4 | 0
  Absolute Neutophil Grade 1-4 | 1
  Absolute Neutophil Grade 4-4 | 0
  Platelet Count Grade 1-4 | 4
  Platelet Count Grade 3-4 | 1
  Hemoglobin Grade 1-4 | 15
  Hemoglobin Grade 3-4 | 2
  Lymphocytes Grade 1-4 | 13
  Lymphocytes Grade 3-4 | 3

5. Secondary Outcome: Number of Participants With Liver Function Laboratory Abnormalities
Description: Abnormal laboratory results were reported after the induction period start and within 90 days after induction period end date. Induction Period was 1 dose every 3 weeks for 4 doses (12 weeks). Common Terminology Criteria (CTC) version 3.0 was used in this study; Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death. Liver Function parameters included: alanine aminotransaminase (ALT), aspartate aminotransferase (AST), Total Bilirubin, and Alkaline Phosphatase (Alk Phos). The most recent assessment on or before Day 1 of study medication was taken as baseline (in addition, baseline laboratory must have been collected no earlier than Day -28).
Time Frame: Baseline to 90 days post last dose, up to July 2014
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
participants
  ALT Grade 1-4 | 11
  ALT Grade 3-4 | 1
  AST Grade 1-4 | 10
  AST Grade 3-4 | 3
  Total Bilirubin Grade 1-4 | 3
  Total Bilirubin Grade 3-4 | 1
  Alk Phos Grade 1-4 | 10
  Alk Phos Grade 3-4 | 1

6. Secondary Outcome: Number of Participants With Renal Laboratory Abnormalities
Description: Abnormal laboratory results were reported after the induction period start and within 90 days after induction period end date. Induction Period was 1 dose every 3 weeks for 4 doses (12 weeks). Common Terminology Criteria (CTC) version 3.0 was used in this study; Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death. Renal parameter=Creatinine. The most recent assessment on or before Day 1 of study medication was taken as baseline (in addition, baseline laboratory must have been collected no earlier than Day -28).
Time Frame: Baseline to 90 days post last dose, up to July 2014
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
participants
  Creatinine Grade 1-4 | 5
  Creatinine Grade 3-4 | 1

7. Secondary Outcome: Number of Participants With Complete Response, Partial Response, Stable Disease, or Progressive Disease as the Best Overall Response
Description: Overall response (OR) was determined using modified World Health Organization (mWHO) criteria. Complete response (CR): complete disappearance of all index and non-index lesions, and no new lesions. Partial response (PR): decrease in index lesions of 50% or greater in a sum of the products of diameters (SPD) relative to baseline, and no new lesions. Stable Disease (SD): Does not meet criteria for CR or PR, in the absence of PD in index lesions and no change or any change with persistence of one or more non-index lesions, and no new lesions. Progressive Disease (PD): At least 25% increase in SPD relative to nadir in index lesions and unequivocal progression of non-index lesions, along with new lesions or no new lesions; or PD: new lesions with any response with index or non-index lesions. Not Evaluable: Response cannot be determined.
Time Frame: Day 1 to 90 days post last dose, up to February 2015 (approximately 2 years)
Population: All participants in the study who received at least one dose of treatment with ipilimumab were summarized.
Measure: Number; unit: participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
participants
  Partial Response (PR) | 2
  Stable Disease (SD) | 2
  Progressive Disease (PD) | 13
  Not Evaluable | 3

8. Secondary Outcome: Percent of Participants With Best Overall Response (BOR) of Complete Response or Partial Response
Description: Best Overall Response Rate (BORR) was defined as the total number of participants whose Best Overall Response (BOR) is Complete Response (CR) or Partial Response (PR) divided by the total number of treated participants (%). A two-sided, exact 95% Confidence Interval (Clopper and Pearson) for the BORR was calculated. Overall response (OR) was determined using modified World Health Organization (mWHO) criteria: Complete Response = complete disappearance of all index and non-index lesions, and no new lesions. Partial Response = decrease in index lesions of 50% or greater in a SPD relative to baseline, and no new lesions. BOR=an overall response of CR or PR at Week 12 or after Week 12.
Time Frame: Day 1 to 90 days post last dose, up to February 2015 (approximately 2 years)
Population: All participants in the study who received at least one dose of treatment with ipilimumab were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 20
percentage of participants | 10.0 [1.2 to 31.7]

ADVERSE EVENTS:
Time Frame: Day 1 to 90 days post last dose, up to February 2015 (approximately 2 years)
Description: Study initiated: December 2013; Study Completion: February 2015
Arm/Group | Ipilimumab
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=20)
C-reactive protein increased (Investigations) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multi-organ failure (General disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Alanine aminotransferase increased (Investigations) | 2
Cerebral infarction (Nervous system disorders) | 1
Erysipelas (Infections and infestations) | 1
Hydrocephalus (Nervous system disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ileus (Gastrointestinal disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=20)
Abdominal pain upper (Gastrointestinal disorders) | 2
Blood bilirubin increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hot flush (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Weight decreased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Headache (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 4
Confusional state (Psychiatric disorders) | 2
Conjunctivitis allergic (Eye disorders) | 1
Delirium (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Haemoglobin decreased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Blood sodium decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Otitis externa (Infections and infestations) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Platelet count decreased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 4
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Oral herpes (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Somnolence (Nervous system disorders) | 2
VIth nerve paralysis (Nervous system disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Erysipelas (Infections and infestations) | 1
Fatigue (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 3
Malaise (General disorders) | 3
Mucosal inflammation (General disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pyrexia (General disorders) | 6
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Urinary retention (Renal and urinary disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Oedema peripheral (General disorders) | 1
Anxiety (Psychiatric disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Cellulitis (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Deep vein thrombosis (Vascular disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.